CLINICAL TRIAL: NCT04605653
Title: Individualized Diet Improvement Program for Weight Loss and Maintenance
Brief Title: Individualized Diet Improvement Program for Weight Loss and Maintenance, Cohort 1
Acronym: iDIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Mindy Lee, Graduate Research Assistant, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18069_cohort1
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Obesity; Overweight; Weight Loss; Diet Habit
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Before and after study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Management Intervention (Experimental): During a 12-month period, participants will attend a total of 22 diet improvement sessions, each of which will last approximately 1 hour. Twelve sessions will be held in the first 5 months and will be focused on safe and efficient weight loss. The participants will learn to create a personalized weight loss diet from their kitchen based on their diet practice and food preference. The next 10 sessions will be held in the last 7 months and will be focused on weight maintenance and healthy eating. The participants will build skills to select foods and create meals that prevent them from overeating.
  Interventions: Behavioral: Weight Management Intervention

INTERVENTIONS:
Behavioral: Weight Management Intervention — Participants attend group and individual dietary education sessions. Participants create a diet plan that satisfies their needs. Participants aim to lose 1 pound weekly until a BMI of 25 is reached. Participants are evaluated through daily self-weighing, dietary records, and food frequency questionnaires.

SUMMARY:
This research is to develop a weight loss and weight maintenance program through dietary modifications for adults with obesity. Although scientific studies have shown the feasibility of rapid and safe dietary weight loss and subsequent weight maintenance, no efficacious dietary weight management program is widely available, and thus bariatric surgery remains the most reliable approach for weight loss/management. Safe and effective dietary weight loss and subsequent weight maintenance require flexible, individualized advice by an experienced dietitian/nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) >28 kg/m2;
* not currently pregnant or lactating;
* have Wi-Fi at home, a working email, and an iPhone or Android smartphone;
* no self-reported severe metabolic, cardiovascular or musculoskeletal disease;
* not using insulin injection;
* able to attend the 22 (1 hour) diet improvement sessions;
* willing to lose 20 lb. or more for 6 months and maintain a healthy weight for one year;
* keep weighing their weight for one and a half years;
* fluent in reading and writing English.

Exclusion Criteria:

* age <18 or >64 years;
* body mass index of <28 kg/m2;
* currently pregnant;
* currently lactating;
* self-reported with severe metabolic, cardiovascular, or musculoskeletal disease;
* use insulin injection;
* not able to attend the 22 (1 hour) diet improvement sessions for 1 year;
* failed to set up a Wi-Fi scale;
* failed to submit a FFQ.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
Body weight | Change from baseline (0 month) to 6 month, 12 month, and 18 month
  Body weight in kilograms measured on a standard scale (Weight Gurus, Greater Goods LLC, MO)

SECONDARY OUTCOMES:
Waist circumference | Change from baseline (0 month) to 12 month
  Waist circumference in centimeters measured using a standard measuring tape
Hip circumference | Change from baseline (0 month) to 12 month
  Hip circumference in centimeters measured using a standard measuring tape
Protein intake | Change from baseline (0 month) to 12 month
  Protein intake in grams and grams/100 kilo-calories using a food frequency questionnaire (FFQ)
Protein intake | Periodically from baseline (0 month) to 12 month
  Protein intake in grams and grams/100 kilo-calories using a 24-hour food record
Fiber intake | Change from baseline (0 month) to 12 month
  Fiber intake in grams and grams/100 kilo-calories using a food frequency questionnaire (FFQ)
Fiber intake | Periodically from baseline (0 month) to 12 month
  Fiber intake in grams and grams/100 kilo-calories using a 24-hour food record

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No